CLINICAL TRIAL: NCT05268978
Title: SHAPES Advanced Telemonitoring of Patients With Heart Failure in Home Environment
Brief Title: Advanced Telemonitoring of Patients With Heart Failure in Home Environment
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Ladislav Stanke, Principal Investigator, University Hospital Olomouc
Other Study IDs: SHAPES UC-PT3-001c
Record Dates: First submitted 2022-01-31; First posted 2022-03-07 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medimonitor — A digital solution consisting of smartphone/tablet based application gathering data from medical and other devices provided to the patients. These devices are as follows: tablet, smartwatch, mobile ECG, blood pressure monitor, weight scales, pulse oximetry device.

SUMMARY:
Heart failure is currently not only a major medical but also a socio-economic problem. Its prevalence is estimated at 1-2% of the population with an exponential increase in older age groups. A very important part of the treatment of heart failure is the gradual uptitration of therapy to the maximum tolerated doses. Properly conducted therapy titration requires more frequent patient contact. Thanks to the introduction of telemedicine techniques, the investigators can communicate more effectively with the patient, reach the target doses of heart failure medication faster and subsequently reduce the number of hospitalizations due to worsening of heart failure.

This study investigates effect of advanced telemonitoring of patients with heart failure in home environment.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤ 40%
* exclusion of obstructive coronary artery disease
* NTproBNP ≥ 125pg/ml
* ≥ 60 years of age
* Informed written and verbal consent
* Able to participate in study activities

Exclusion Criteria:

* LVEF ≥ 40%
* Ischaemic ethiology of cardiomyopathy
* NTproBNP ≤ 125pg/ml
* Severe psychological disturbances
* Absence of collaboration (informed consent)
* BP ≤ 110mmHg without hypertensive medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed heart failure with reduced ejection fraction due to non-ischemic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of step telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from the medical and other devices (tablet with smartwatch providing data from the pedometer, i.e. number of steps) provided to the patients with heart failure in home environment.
Evaluation of the effect of ECG telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from medical and other devices (tablet with mobile ECG) provided to the patients with heart failure in home environment.
Evaluation of the effect of blood pressure telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from medical and other devices (tablet and blood pressure monitor recording systolic and diastolic blood pressure) provided to the patients with heart failure in home environment.
Evaluation of the effect of body weight telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from medical and other devices (tablet and diagnostic weight scales for monitoring weight in kilograms) provided to the patients with heart failure in home environment.
Evaluation of the effect of body water telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from medical and other devices (tablet and diagnostic weight scales for monitoring body water percentage) provided to the patients with heart failure in home environment.
Evaluation of the effect of blood oxygen saturation telemonitoring during uptitration of heart failure medication. | 3 month
  Uptitration of therapy guided by data from medical and other devices (tablet and pulse oximetry device to monitor blood oxygen saturation in percents) provided to the patients with heart failure in home environment.
Evaluation of changes of NTproBNP levels at the beginning vs. at the end of the study. | 3 month
  Evaluation of changes of NTproBNPlevels as a marker of effective therapy of heart failure.
Evaluation of changes in LVEF echocardiographic parameter at the beginning vs. at the end of study. | 3 month
  Assessment of the effect of heart failure therapy (left ventricular reverse remodelation) by evaluation of changes in LVEF echocardiographic parameter
Evaluation of changes in LVEDD echocardiographic parameter at the beginning vs. at the end of study. | 3 month
  Assessment of the effect of heart failure therapy (left ventricular reverse remodelation) by evaluation of changes in LVEDD echocardiographic parameter
Evaluation of changes in LVESD echocardiographic parameter at the beginning vs. at the end of study. | 3 month
  Assessment of the effect of heart failure therapy (left ventricular reverse remodelation) by evaluation of changes in LVESD echocardiographic parameter
Evaluation of changes in LAVi echocardiographic parameter at the beginning vs. at the end of study. | 3 month
  Assessment of the effect of heart failure therapy (left ventricular reverse remodelation) by evaluation of changes in LAVi echocardiographic parameter
Evaluation of changes in diastolic dysfunction by echocardiography at the beginning vs. at the end of study. | 3 month
  Assessment of the effect of heart failure therapy (left ventricular reverse remodelation) by evaluation of changes in diastolic dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine I - Cardiology, University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No